CLINICAL TRIAL: NCT00441714
Title: Effect of Ischemic Postconditioning on Targeting of Annexin A5 After Forearm Exercise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: new insights have let us to expect marginal annexin targeting with a 10 minutes delay between reperfusion and administration of Annexin A5
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: IPost
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Cardiovascular Disease; Ischemia-reperfusion Injury; Postconditioning
Keywords: cardiovascular disease; ischemia-reperfusion injury; postconditioning; annexin targeting
MeSH Terms: conditions — Cardiovascular Diseases; Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: repetitive short ischemia and reperfusion of non dominant fore arm after 10 minute ischemic exercise

SUMMARY:
To adjust our forearm model for ischemia reperfusion injury, in order to used it for assessment of ischemia reperfusion damage in elderly and patients.

To test the effect of ischemic postconditioning on ischemia reperfusion injury in healthy volunteers, using Annexin binding after repetitive handgripping.

DETAILED DESCRIPTION:
Recently, ischemic postconditioning has been identified as a protective intervention against ischemia-reperfusion injury. In animal studies, the signalling pathway of this (impressive) protective phenomenon is very similar to ischemic preconditioning. It opens a new avenue of post-reperfusion interventions with drugs that have been shown to mimic ischemic preconditioning. Before we can study this phenomenon in our forearm ischemia-reperfusion model, we need additional validating experiments. The purpose of this study proposal is to provide these data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* No physical limitation to perform ischemic exercise
* Informed consent

Exclusion Criteria:

* Diabetes (fasting glucose > 7,0mmol/l, or random glucose >11,0mmol/l)
* hyperlipidemia (random total cholesterol > 6.5 mmol/l)
* Hypertension (supine SBP/DBP > 140/90 mmHg at screening)
* Any cardiovascular disease
* Drug abuse
* Concomitant chronic use of medication
* Administration of radioactivity in research setting during the last 5 years
* Participation to any drug-investigation during the previous month as checked with VIP check according to CRCN standard procedures.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Annexin A 5 targeting in the non dominant thenar muscle after (ischemic exercise), as a indicator for ischemia reperfusion injury.

SECONDARY OUTCOMES:
Workload during (ischemic) exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD PhD, Principal Investigator — RUMCN
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Background] Rongen GA, Oyen WJ, Ramakers BP, Riksen NP, Boerman OC, Steinmetz N, Smits P. Annexin A5 scintigraphy of forearm as a novel in vivo model of skeletal muscle preconditioning in humans. Circulation. 2005 Jan 18;111(2):173-8. doi: 10.1161/01.CIR.0000151612.02223.F2. Epub 2004 Dec 27. PMID 15623546